CLINICAL TRIAL: NCT03915223
Title: Interest of Preoperative Corticosteroid Therapy for Surgical Fractures of the Lower Limb
Brief Title: Soft Part Management for Surgical Fractures of the Lower Limb
Acronym: ICOMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBHP 2018 BOISGARD; 2018-003565-33 (Other: 2018-003565-33)
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Leg Injuries; Fracture; Edema
Keywords: preoperative procedure; leg fractures; osteosynthesis; corticosteroids
MeSH Terms: conditions — Leg Injuries; Fractures, Bone; Edema

STUDY DESIGN:
Intervention Model Description: Solumedrol (steroidal anti-inflammatory drug) injection
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm "Injection corticosteroids" (Experimental): Single dose of Solumedrol 2 mg/kg
  Interventions: Procedure: leg fracture
- Arm " injection physiological serum" (Placebo Comparator): Single dose of physilogical serum
  Interventions: Procedure: leg fracture

INTERVENTIONS:
Procedure: leg fracture — Surgical leg fracture with injection of solumedrol (steroidal anti-inflammatory drug) or physiological serum

SUMMARY:
The assessment consists in comparing corticoids injection versus placebo in surgery of lower limb fractures The aim of study is to assess (state cutaneous, efficacy, safety) corticoids injection on a prospective, randomized analysis

DETAILED DESCRIPTION:
One of the major problems of below-knee fractures is edema (delaying surgery time and post-operative complications for healing).

The effect corticosteroids (anti-edema and anti-inflammatory) is used in neurosurgery and maxillofacial surgery.

So, it seemed judicious to evaluate the effectiveness of corticosteroids in bolus preoperatively in order to limit the importance of the edema before intervention to prevent adverse effect of the edema on the cicatrization.

This study will aim to confirm this indication or not on the contrary to change current practices.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18, hospitalized in the Orthopedics Department for a leg fracture (ankle, tibia: proximal, diaphysis, distal) requiring surgery within 72 hours of the trauma
* Patient covered by the social security system
* Patient giving informed consent

Exclusion Criteria:

* Open fracture with infectious risks cauchoix 2 and 3
* Multiple trauma,
* Pathological fracture on primary or secondary lesions,
* Pre-existing bone disease (excluding osteoporosis) of the operated limb,
* Diabetes,
* Pre-existing trophic disorders on one of the 2 lower limbs,
* Long-term corticotherapy,
* Pathology of the pituitary-adrenal axis,
* Any other contraindication to glucocorticoids: any infectious condition, some developing viral diseases (including hepatitis, herpes, chicken pox, shingles), hypersensitivity to one of the constituents
* Hypernatremia and hypochloremia
* Pre-existing severe cardiac injury
* Contraindication to TegadermTM
* Patient placed under guardianship, tutorship or safeguard of justice,
* Pregnant or lactating women,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
leg perimeter | 2 days
  measure of leg perimeter at the fractured area compared to the contralateral side

SECONDARY OUTCOMES:
leg perimeter | 15 days
  measure of leg perimeter at the fractured area compared to the contralateral side
leg perimeter | 7 days
  measure of leg perimeter at the fractured area compared to the contralateral side
pain leg | preoperative
  THE VISUAL SIMILAR SCALE is auto-completed. For the intensity of pain, the scale varies between " no pain " (the score of 0) and " the pain so badly as he could be " or " the worst conceivable pain " (the score of 10)
pain leg | 2 days
  THE VISUAL SIMILAR SCALE is auto-completed. For the intensity of pain, the scale varies between " no pain " (the score of 0) and " the pain so badly as he could be " or " the worst conceivable pain " (the score of 10)
pain leg | 7 days
  THE VISUAL SIMILAR SCALE is auto-completed. For the intensity of pain, the scale varies between " no pain " (the score of 0) and " the pain so badly as he could be " or " the worst conceivable pain " (the score of 10)
pain leg | 15 days
  THE VISUAL SIMILAR SCALE is auto-completed. For the intensity of pain, the scale varies between " no pain " (the score of 0) and " the pain so badly as he could be " or " the worst conceivable pain " (the score of 10)
pain leg | 45 days
  THE VISUAL SIMILAR SCALE is auto-completed. For the intensity of pain, the scale varies between " no pain " (the score of 0) and " the pain so badly as he could be " or " the worst conceivable pain " (the score of 10)
pain leg | 3 months
  THE VISUAL SIMILAR SCALE is auto-completed. For the intensity of pain, the scale varies between " no pain " (the score of 0) and " the pain so badly as he could be " or " the worst conceivable pain " (the score of 10)
pain leg | 6 months
  THE VISUAL SIMILAR SCALE is auto-completed. For the intensity of pain, the scale varies between " no pain " (the score of 0) and " the pain so badly as he could be " or " the worst conceivable pain " (the score of 10)
State cutaneous | 7 days
  index form of follow-up the state cutaneous of the wound
State cutaneous | 15 days
  index form of follow-up the state cutaneous of the wound
Lower limb functional scale (EFMI) | 6 months
  The Lower limb functional scale grading system uses 100 points to assess pain, function and mobility of the leg. The score varies between 0 and 100, more the value is better brought up is the score
Complications | 6 months
  list of the complications : Phlyctenes, scar disunity, cutaneous necrosis, infection, phlebitis, compartment syndrome, complex regional pain syndrome, delay of bone consolidation

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Boisgard, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France